CLINICAL TRIAL: NCT02543359
Title: A Statewide Trial to Compare Three Training Models for Implementing an EBT
Brief Title: A Statewide Trial to Compare Three Training Models for Implementing an Evidence-based Treatment (EBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy Herschell, Associate Professor of Psychiatry and Psychology, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO12060529; 5R01MH095750-02 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-09-07 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Training of Mental Health Professionals; Disruptive Behavior Disorders
Keywords: Training; Implementation; Community-Based Mental Health Services; Parent-Child Interaction Therapy; Children
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clinicians and Supervisors (Experimental): After randomization clinicians and supervisors from community behavioral health agencies receive training in one of three PCIT training models: Train the Trainer (TTT), Learning Collaborative (LC) or Web-Supported Self Study (SS).
  Interventions: Behavioral: Training Models of PCIT
- Administrators (Experimental): After randomization administrators from participating community behavioral health agencies receive one of three treatments for PCIT (1/3 Learning Collaborative, 1/3 other treatment - none, and 1/3 other treatment - none).
  Interventions: Behavioral: Training Models of PCIT
- Parent-Child Dyads (Experimental): Parent-child dyads receive Parent-Child Interaction Therapy (PCIT) treatment from trained clinicians/supervisors.
  Interventions: Behavioral: Parent-Child Interaction Therapy (PCIT) Treatment

INTERVENTIONS:
Behavioral: Training Models of PCIT — Agency participants are trained in one of three training model strategies: Train the Trainer Model (TTT), Learning Collaborative (LC), or Web-Supported Self Study (SS).One third of participating agencies will be randomized to the Train the Trainer training model.One third of participating agencies will be randomized to the Learning Collaborative training model.One third of participating agencies will be randomized to the Web-Supported Self Study.
  Arms: Clinicians and Supervisors
Behavioral: Training Models of PCIT — One-third of administrators are trained in the Learning Collaborative training model. One-third of administrators will be trained to usual treatment (none). One-third of administrators will be trained to usual treatment (none).
  Arms: Administrators
Behavioral: Parent-Child Interaction Therapy (PCIT) Treatment — Parent-Child Interaction Therapy (PCIT), a parent coaching evidence-based protocol is given to each family from clinicians and supervisors in each training model.
  Arms: Parent-Child Dyads

SUMMARY:
Evidence-based treatments (EBTs) are available for treating Disruptive Behavior Disorders ( DBDs) including Parent-Child Interaction Therapy (PCIT). Despite EBTs' potential to help children and families, they have primarily remained in university settings. Recognized field leaders have expressed concern over the discrepancy between treatment research and clinical practice, and have indicated that EBT implementation is a priority. Little empirical evidence exists regarding how effective commonly used training models are in changing clinician behavior, achieving full implementation (e.g., increasing treatment fidelity, integrating into service settings), and supporting positive client outcomes. This novel application will evaluate the effectiveness of three training models (Learning Collaborative, Train-the-Trainer, and Web-Supported Self-Study) to implement a well-established EBT in real-world, community settings.

To accomplish this goal, the project will be guided by three specific aims:

1. to build knowledge about training outcomes,
2. to build knowledge about implementation outcomes, and
3. to understand the impact of training clinicians using LC, TTT, and SS models on key client outcomes.

Seventy-two of 243 possible (30%) licensed psychiatric clinics across Pennsylvania will be randomized to one of three training conditions:

1. Learning Collaborative (LC),
2. Train-the-Trainer (TTT), or
3. Web-Supported Self-Study (SS).

Data also will be collected on staff trained by clinicians in the TTT group given that the intention of a TTT model is for participants of that group to return to their organization and train others within the organization. The impact of training (clinician level) will be evaluated at 4 time-points coinciding with the training schedule: baseline, 6, 12, and 24-months. Immediately after training begins, parent-child dyads (client level) will be recruited from the caseloads of participating clinicians (N = 288). Client outcomes will be assessed at four timepoints (pre-treatment, 3, 6, and 12-months). Implementation outcomes (clinic level) will be assessed at baseline, 6, 12, and 24-months after training. This proposal builds on an ongoing state-led initiative to implement, and ultimately sustain, PCIT statewide. Lessons learned from this project will directly impact future EBT implementation efforts in Pennsylvania and other states, helping to increase the use of EBTs in community settings nationwide.

ELIGIBILITY:
Inclusion Criteria:

Administrators group

* must be employed at an agency selected to participate in training as an Executive Director, Chief Financial Officer, or other person responsible for daily operations.

Clinicians/Supervisors group

* a masters or doctoral level professional in the human services field (e.g., social work, psychology, education),
* licensed in his/her field or receiving supervision from a licensed individual,
* actively seeing children and families who are appropriate for PCIT,
* receptive to training in PCIT but not previously trained in PCIT,
* amenable to study tasks (e.g., video-taping, completing assessments).

Parent-Child Dyads group

* Any parent-child dyad who a trained clinician enrolls in PCIT services

Exclusion Criteria:

Administrators group

* not employed at an agency selected to participate in training as an Executive Director, Chief Financial Officer, or other person responsible for daily operations.

Clinicians group

* a bachelors or lower level professional in the human services field,
* unlicensed in his/her field or not receiving supervision from a licensed individual,
* not actively seeing children and families who are appropriate for PCIT,
* not receptive to training in PCIT but not previously trained in PCIT, and/or
* not amenable to study tasks. Interns also will be excluded.

Parent-Child Dyads group

- if he/she is a ward of the state or living in state custody

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2012-09; Primary Completion 2017-11-02 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Clinician knowledge of treatment based on PCIT Coaches Quiz | Measured at baseline, 6, 12, and 24 months
  The PCIT Coaches Quiz measures clinicians' knowledge of PCIT concepts; a scale to assess clinicians' knowledge of PCIT concepts and coaching scenarios, and is a mixed question format of multiple choice and short answer. It was created by PCIT Developers based on training content.
Change in Clinician PCIT skill competency based on Therapist Competency Checklist | Measured at baseline and 6, 12, and 24 months
  Therapist Competency Checklist evaluates competency criteria based on established Training Guidelines. The criteria are divided into five categories representing the full PCIT protocol (e.g., assessment, treatment, coaching). These pre-determined, skill-based competency items are rated by the trainer after observing trainees behavior over 1 year.
Change in Clinician attitudes about training based on Feedback Surveys | Measured at baseline and 6, 12 months and 24 months
  The following areas are measured: satisfaction with implementation condition,treatment acceptability,understanding, feasibility, and systems support; and satisfaction with training content, format, and presenters.

SECONDARY OUTCOMES:
Change in PCIT administrative interviews | Measured at baseline and 6, 12 months and 24 months
  Agency acceptability, adoption, appropriateness, cost feasibility, fidelity, penetration and sustainability of PCIT.
Change in PCIT patient functioning | Measured at baseline, 3, 6 and 12 months
  Family Outcome - Client mental health functioning (symptom improvement and daily functioning), treatment satisfaction, barriers to treatment, and service use (additional services and PCIT treatment process).

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Herschell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Jackson CB, Macphee FL, Hunter LJ, Herschell AD, Carter MJ. Enrolling Family Participants in a Statewide Implementation Trial of an Evidence-Based Treatment. Prog Community Health Partnersh. 2017;11(3):233-241. doi: 10.1353/cpr.2017.0028. PMID 29056615
- [Background] Herschell AD, Scudder AB, Schaffner KF, Slagel LA. Feasibility and Effectiveness of Parent-Child Interaction Therapy with Victims of Domestic Violence: A Pilot Study. J Child Fam Stud. 2017 Jan;26(1):271-283. doi: 10.1007/s10826-016-0546-y. Epub 2016 Sep 19. PMID 28503060
- [Background] Herschell AD, Kolko DJ, Scudder AT, Taber-Thomas S, Schaffner KF, Hiegel SA, Iyengar S, Chaffin M, Mrozowski S. Protocol for a statewide randomized controlled trial to compare three training models for implementing an evidence-based treatment. Implement Sci. 2015 Sep 28;10:133. doi: 10.1186/s13012-015-0324-z. PMID 26416029
- [Background] Scudder AT, Taber-Thomas SM, Schaffner K, Pemberton JR, Hunter L, Herschell AD. A mixed-methods study of system-level sustainability of evidence-based practices in 12 large-scale implementation initiatives. Health Res Policy Syst. 2017 Dec 7;15(1):102. doi: 10.1186/s12961-017-0230-8. PMID 29216886
- [Derived] Herschell AD, Kolko DJ, Scudder AT, Taber-Thomas SM, Schaffner KF, Hart JA, Mrozowski SJ, Hiegel SA, Iyengar S, Metzger A, Jackson CB. A Statewide Randomized Controlled Trial to Compare Three Models for Implementing Parent Child Interaction Therapy. J Clin Child Adolesc Psychol. 2023 Nov-Dec;52(6):780-796. doi: 10.1080/15374416.2021.2001745. Epub 2021 Dec 20. PMID 34928748